CLINICAL TRIAL: NCT01436370
Title: A Phase II Study in Adults With Rheumatoid Arthritis Receiving TNF-alpha-inhibitor Therapy to Assess the Immunogenicity and Safety of Trivalent Inactivated Vaccine (TIV) and High Dose Trivalent Inactivated Vaccine (High-Dose TIV) Administered at Two Dosage Levels
Brief Title: TIV and High Dose TIV in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10-0076
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2013-02

CONDITIONS: Influenza
Keywords: influenza, rheumatoid arthritis, TNF-alpha-inhibitor, Fluzone®, Fluzone® High Dose
MeSH Terms: conditions — Influenza, Human; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Group 1 Controls (Experimental): 40 (up to 50) adults, healthy gender and age-matched controls, given a single 15 mcg intramuscular dose of Sanofi Pasteur Fluzone®
  Interventions: Biological: Trivalent inactivated influenza vaccine
- Group 2 (Experimental): 40 (up to 50) adults with Rheumatoid Arthritis receiving TNF-alpha-inhibitor therapy, given a single 60 mcg intramuscular dose of Sanofi Pasteur Fluzone® High Dose.
  Interventions: Biological: Trivalent inactivated influenza vaccine
- Group 2 Controls (Experimental): 40 (up to 50) adults, healthy gender and age-matched controls, given a single 60 mcg intramuscular dose of Sanofi Pasteur Fluzone® High Dose.
  Interventions: Biological: Trivalent inactivated influenza vaccine
- Group 1 (Experimental): 40 (up to 50) adults with Rheumatoid Arthritis receiving TNF-alpha-inhibitor therapy, given a single 15 mcg intramuscular dose of Sanofi Pasteur Fluzone®
  Interventions: Biological: Trivalent inactivated influenza vaccine

INTERVENTIONS:
Biological: Trivalent inactivated influenza vaccine — Inactivated trivalent influenza virus vaccine (Sanofi Pasteur Fluzone® High Dose [60 mcg x 3 strains]), as a single intramuscular dose. 80 and up to 100 subjects. Subjects enrolling between October 2011 and February 2012 will receive the 2011-2012 vaccine and subjects enrolling after July 2012 will receive the 2012-2013 vaccine.
  Arms: Group 2; Group 2 Controls
Biological: Trivalent inactivated influenza vaccine — Inactivated trivalent influenza virus vaccine (Sanofi Pasteur Fluzone® [15 mcg x 3 strains]), as a single intramuscular dose. 80 and up to 100 subjects. Subjects enrolling between October 2011 and February 2012 will receive the 2011-2012 vaccine and subjects enrolling after July 2012 will receive the 2012-2013 vaccine.
  Arms: Group 1; Group 1 Controls

SUMMARY:
A randomized, double-blinded, Phase II study in adults with Rheumatoid Arthritis receiving TNF-alpha-inhibitor therapy aged 18 to 64 years of age and healthy gender-and age-matched control subjects . This study will investigate the immunogenicity, safety, and reactogenicity of two different doses of inactivated trivalent influenza virus vaccine (Sanofi Pasteur Fluzone [15 mcg x 3 strains] and Sanofi Pasteur Fluzone High Dose [60 mcg x 3 strains]) administered intramuscularly in individuals with rheumatoid arthritis receiving anti-TNF-alpha (TNFi) therapy and healthy age- and gender- matched controls.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, Phase II study in adults with Rheumatoid Arthritis receiving TNF-alpha inhibitor therapy, aged 18 years to 64 years of age. This study is designed to investigate the immunogenicity, safety, and reactogenicity of two different doses of inactivated trivalent influenza virus vaccine given at two dose levels (15 mcg and 60 mcg) administered IM in individuals with rheumatoid arthritis receiving anti-TNF-alpha therapy or age and gender matched control subjects. The study is conducted over two seasons, 2011-2012 and 2012-2013. Subjects enrolling between October 2011 and February 2012 will receive the 2011-2012 vaccine, while those enrolling after July 2012 will receive the 2012-2013 vaccine. Immunogenicity testing will determine the proportion of subjects in each group with titer a 4-fold rise in HAI titers (defined as either a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer >/=1:40 or a pre-vaccination HAI titer >/=1:10 and a minimum four-fold rise in post-vaccination HAI titer) against each of the specific influenza strains included in vaccine the subject received at day 21 following vaccination. The proportion of subjects in each group achieving a serum HAI titer of >/= 1:40 or a 4-fold rise in HAI titer or greater in HAI titer against each strain in the vaccine compared to the controls subjects. Safety testing will assess the occurrence of vaccine-associated Serious adverse events (SAEs) throughout the course of the study, and the occurrence of solicited local and systemic adverse events (AEs) within 8 days post vaccination. Solicited AEs (including rheumatoid arthritis clinical status) will be assessed during the course of the study. Subjects will have four face to face visits and one telephone contact. Day 0 will include the consent process, a medical history and physical exam for the RA subjects to assess the activity of their RA at the time of enrollment, vital signs, phlebotomy for prevaccine serology. Subjects will be randomized to receive IM seasonal TIV or High-Dose TIV at this visit and will receive the assigned vaccine. They will be observed for 20 minutes and will be taught to fill out a 7 day memory aid that will assess daily temperature, local and systemic reactogenicity. A telephone call will be made to assess reactogenicity and to review the memory aid on day 3. Subjects will return on day 7 for review of the memory aid, AEs/SAEs, vital signs and phlebotomy for serology. A physical exam will be performed if indicated. They will return on day 21 and at 6 months for review of AEs/SAEs, vital signs and phlebotomy for serology. A physical exam will be performed if indicated.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for RA Subjects

* Male or non-pregnant female between the ages of 18 and 64 years, inclusive, who has stable RA and has received TNFi therapy during the previous 3 months.
* Female subjects: for the 30 days prior to enrollment through 30 days following receipt of TIV or HTIV vaccine must fulfill one of the following: (i) she is not able to bear children because she has been surgically sterilized (tubal ligation or hysterectomy) for at least one year or is at least 1 year post-menopausal or (ii) she agrees to practice effective methods of contraception including, but not limited to, abstinence, barrier methods (such as a condom or diaphragm) used with a spermicide, birth control pills, patches or hormonal shots or hormonal implants, NuvaRing and IUDs (intrauterine devices). Adherence to contraceptive method will be captured on the appropriate case report form (CRF).
* In good health, as determined by vital signs (see toxicity table in section 9.2.1.1), medical history to ensure any existing medical diagnoses or conditions are stable and not considered clinically significant, and physical examination.
* Intend to be available through 6 months following receipt of vaccine.
* Able to understand and comply with planned study procedures.
* Provide written informed consent prior to initiation of any study procedures.

Inclusion Criteria for Healthy Subjects

* Male or non-pregnant female between the ages of 18 and 64 years, inclusive.
* Female subjects: for the 30 days prior to enrollment through 30 days following receipt of TIV or HTIV vaccine must fulfill one of the following: (i) she is not able to bear children because she has been surgically sterilized (tubal ligation or hysterectomy) for at least one year or is at least 1 year post-menopausal or (ii) she agrees to practice effective methods of contraception including, but not limited to, abstinence, barrier methods (such as a condom or diaphragm) used with a spermicide, birth control pills, patches or hormonal shots or hormonal implants, NuvaRing and IUDs (intrauterine devices). Adherence to contraceptive method will be captured on the appropriate case report form (CRF).
* In good health, as determined by vital signs (see toxicity table in section 9.2.1.1), medical history to ensure any existing medical diagnoses or conditions are stable and not considered clinically significant, and physical examination.
* Intend to be available through 6 months following receipt of vaccine.
* Able to understand and comply with planned study procedures.
* Provide written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

Exclusion Criteria for all Subjects

* For subjects enrolled after July 2012: Enrolled in this study during the 2011-2012 flu season.
* Has received the seasonal influenza vaccine for the current season. For subjects enrolling between October 2011 and February 2012, this is the 2011-2012 seasonal influenza vaccine. For subjects enrolling after July 2012, this is the 2012-2013 seasonal influenza vaccine.
* Has a known allergy to eggs, egg proteins or other components in the vaccines (i.e. formaldehyde, gelatin sodium phosphate, sodium chloride, octylphenol ethoxylate).
* Has a known or suspected latex allergy or sensitivity.
* Has a positive urine or serum pregnancy test within 24 hours prior to vaccination (if female of childbearing potential as defined in Inclusion criterion 2), or women who are breastfeeding.
* Has a history of severe reactions following immunization with contemporary influenza virus vaccines.
* Has an active neoplastic disease or a history of any hematologic malignancy (cancers of blood or bone marrow) or current bleeding or blood clotting disorder.
* For "healthy volunteer" (without RA) subjects: Long term (at least 14 days of prednisone 2 mg/kg or equivalent other glucocorticoid) use of oral, parenteral or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months. (Nasal and topical steroids are allowed.)
* Has a diagnosis of a current and uncontrolled major psychiatric disorder.
* Has been hospitalized in the past 10 years for psychiatric illness, suicide attempt, or confinement for danger to self or others.
* Is receiving listed psychiatric drugs as below*. Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment, without decompensating are allowed enrollment into the study.

  * aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, trifluopromazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate, lithium citrate, lamotrigine, prochlorperazine, paliperidone or iloperidone.
* Has a history of receiving immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
* Has received an experimental/investigational agent (vaccine, drug, biologic, device, blood product, or medication) within 28 days prior to vaccination in this study, or expects to receive an experimental/investigational agent within the study time period (180 days after vaccination in this study).
* Is participating or plans to participate in another clinical trial with a licensed product during the 6-month study period.
* Has received any other licensed vaccines within 14 days (for inactivated vaccines) or 21 days (for live vaccines) prior to vaccination in this study, or expects to receive a licensed vaccine during the 21 days after vaccination in this study.
* Has received antiviral agent against influenza A and/or B within 48 hours prior to vaccination in this study. Antiviral agents should not be administered until 2 weeks after vaccination in this study unless medically necessary.
* Has an acute or chronic medical condition other than RA that, in the opinion of the investigator, would interfere with the evaluation of responses (this includes, but is not limited to: known chronic liver, lung or heart disease, chronic anemia, (non-RA subjects only), metabolic disorders such as diabetes (resolved gestational diabetes is acceptable), significant renal disease, transplant recipients, system lupus erythematosus, psoriatic arthritis or gout).
* Has a moderate to severe acute illness and/or an oral temperature greater than or equal to 100.4 degrees Fahrenheit, within 72 hours prior to vaccination. (This may result in a temporary delay of vaccination).
* Immunosuppression as a result of an underlying illness or treatment other than RA therapy, or use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months.
* Known infection with HIV, Hepatitis B or Hepatitis C infection or autoimmune hepatitis.
* Has a history of alcohol or drug abuse in the last 5 years.
* Has a history of Guillain-Barré Syndrome.
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa - Vaccine Research & Education Unit, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults with rheumatoid arthritis (RA) receiving tumor necrosis factor (TNF)-alpha-inhibitor therapy and healthy controls were recruited from existing volunteer populations and the community around the clinical site. Participants were enrolled between 20OCT2011 - 3JAN2012 (2011-2012 vaccine); and 12SEP2012 -14JAN2013 (2012-2013 vaccine).
Groups:
- RA Participants, 2011-2012 Fluzone Standard Dose: Adults with Rheumatoid Arthritis receiving TNF-alpha-inhibitor therapy were given a single 15 mcg intramuscular dose of 2011-2012 Sanofi Pasteur Fluzone®
- Healthy Controls, 2011-2012 Fluzone Standard Dose: Healthy gender and age-matched controls were given a single 15 mcg intramuscular dose of 2011-2012 Sanofi Pasteur Fluzone®
- RA Participants, 2011-2012 Fluzone High Dose: Adults with Rheumatoid Arthritis receiving TNF-alpha-inhibitor therapy were given a single 60 mcg intramuscular dose of 2011-2012 Sanofi Pasteur Fluzone® High Dose
- Healthy Controls, 2011-2012 Fluzone High Dose: Healthy gender and age-matched controls were given a single 60 mcg intramuscular dose of 2011-2012 Sanofi Pasteur Fluzone® High Dose
- RA Participants, 2012-2013 Fluzone Standard Dose: Adults with Rheumatoid Arthritis receiving TNF-alpha-inhibitor therapy were given a single 15 mcg intramuscular dose of 2012-2013 Sanofi Pasteur Fluzone®
- Healthy Controls, 2012-2013 Fluzone Standard Dose: Healthy gender and age-matched controls were given a single 15 mcg intramuscular dose of 2012-2013 Sanofi Pasteur Fluzone®
- RA Participants, 2012-2013 Fluzone High Dose: Adults with Rheumatoid Arthritis receiving TNF-alpha-inhibitor therapy were given a single 60 mcg intramuscular dose of 2012-2013 Sanofi Pasteur Fluzone® High Dose
- Healthy Controls, 2012-2013 Fluzone High Dose: Healthy gender and age-matched controls were given a single 60 mcg intramuscular dose of 2012-2013 Sanofi Pasteur Fluzone® High Dose
Period: Overall Study
Arm/Group | RA Participants, 2011-2012 Fluzone Standard Dose | Healthy Controls, 2011-2012 Fluzone Standard Dose | RA Participants, 2011-2012 Fluzone High Dose | Healthy Controls, 2011-2012 Fluzone High Dose | RA Participants, 2012-2013 Fluzone Standard Dose | Healthy Controls, 2012-2013 Fluzone Standard Dose | RA Participants, 2012-2013 Fluzone High Dose | Healthy Controls, 2012-2013 Fluzone High Dose
Started | 6 | 6 | 10 | 10 | 19 | 19 | 16 | 16
Completed | 6 | 6 | 10 | 10 | 18 | 19 | 16 | 16
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants who were enrolled and vaccinated.
Groups:
- Total: Total of all reporting groups
Arm/Group | RA Participants, 2011-2012 Fluzone Standard Dose | Healthy Controls, 2011-2012 Fluzone Standard Dose | RA Participants, 2011-2012 Fluzone High Dose | Healthy Controls, 2011-2012 Fluzone High Dose | RA Participants, 2012-2013 Fluzone Standard Dose | Healthy Controls, 2012-2013 Fluzone Standard Dose | RA Participants, 2012-2013 Fluzone High Dose | Healthy Controls, 2012-2013 Fluzone High Dose | Total
Number analyzed (Participants) | 6 | 6 | 10 | 10 | 19 | 19 | 16 | 16 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (9.3) | 46.4 (9.4) | 47.6 (9.5) | 48.3 (10.1) | 49.8 (11.0) | 50.1 (10.8) | 52.8 (9.5) | 52.1 (9.4) | 49.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 7 | 7 | 11 | 11 | 9 | 9 | 64
  Male | 1 | 1 | 3 | 3 | 8 | 8 | 7 | 7 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 6 | 5 | 10 | 7 | 19 | 18 | 15 | 15 | 95
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 5 | 6 | 10 | 10 | 18 | 19 | 15 | 16 | 99
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 10 | 10 | 19 | 19 | 16 | 16 | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of RA Participants in the 2011-2012 Season Who Achieved Seroconversion at Day 21 Against Each of the 3 Specific Influenza Strains in Vaccine the Participant Received
Description: Blood was collected from RA participants prior to vaccination and at the 21 day follow up visit for testing in the HAI assay with 2011-2012 seasonal influenza vaccine strains virus as the assay antigens. A participant met the threshold of seroconversion if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to and Day 21 following immunization
Population: The analysis population includes all RA participants enrolled and vaccinated with the 2011-2012 vaccines.
Measure: Number; unit: participants
Arm/Group | RA Participants, 2011-2012 Fluzone Standard Dose | RA Participants, 2011-2012 Fluzone High Dose
Number analyzed (Participants) | 6 | 10
participants
  B/Brisbane/60/2008 | 1 | 6
  A/Perth/16/2009 (A/H3N2) | 1 | 6
  A/California/7/2009 (A/H1N1) | 4 | 7
Statistical Analysis 1: Comparison: RA Participants, 2011-2012 Fluzone Standard Dose vs RA Participants, 2011-2012 Fluzone High Dose; This is the comparison for the B/Brisbane/60/2008 strain; Test type: Superiority or Other; p = 0.145, Fisher Exact
Statistical Analysis 2: Comparison: RA Participants, 2011-2012 Fluzone Standard Dose vs RA Participants, 2011-2012 Fluzone High Dose; This is the comparison for the A/Perth/16/2009 (A/H3N2) strain; Test type: Superiority or Other; p = 0.145, Fisher Exact
Statistical Analysis 3: Comparison: RA Participants, 2011-2012 Fluzone Standard Dose vs RA Participants, 2011-2012 Fluzone High Dose; This is the comparison for the A/California/7/2009 (A/H1N1) strain; Test type: Superiority or Other; p = 0.999, Fisher Exact

2. Secondary Outcome: Number of Participants Reporting Vaccine-related Serious Adverse Events (SAEs) Throughout the Course of the Study.
Description: Serious adverse events included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required in-patient hospitalization or prolongation thereof; resulted in a congenital anomaly/birth defect; or may have jeopardized the participant or required intervention to prevent one of these outcomes. Association to vaccination was determined by a study clinician licensed to make medical diagnosis.
Time Frame: Day 0 to Day 180
Population: The analysis population includes all participants enrolled and vaccinated in the study.
Measure: Number; unit: participants
Arm/Group | RA Participants, 2011-2012 Fluzone Standard Dose | Healthy Controls, 2011-2012 Fluzone Standard Dose | RA Participants, 2011-2012 Fluzone High Dose | Healthy Controls, 2011-2012 Fluzone High Dose | RA Participants, 2012-2013 Fluzone Standard Dose | Healthy Controls, 2012-2013 Fluzone Standard Dose | RA Participants, 2012-2013 Fluzone High Dose | Healthy Controls, 2012-2013 Fluzone High Dose
Number analyzed (Participants) | 6 | 6 | 10 | 10 | 19 | 19 | 16 | 16
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Geometric Mean Titers (GMT) for Each of the Specific Influenza Strains Included in Vaccine Received by Participants in the 2011-2012 Season
Description: Blood was collected for HAI assay at Day 0 prior to vaccination and again at 7, 21 and 180 days following vaccination. The HAI assay was conducted with the three antigens in the 2011-2012 seasonal inactivated TIV. Within each 2011-2012 study arm, geometric mean titers and 95% confidence intervals were calculated for each antigen separately.
Time Frame: Days 0, 7, 21 and 180
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RA Participants, 2011-2012 Fluzone Standard Dose | Healthy Controls, 2011-2012 Fluzone Standard Dose | RA Participants, 2011-2012 Fluzone High Dose | Healthy Controls, 2011-2012 Fluzone High Dose
Number analyzed (Participants) | 6 | 6 | 10 | 10
titers
  B/Brisbane/60/2008 - Day 0 | 22.4 [7.7 to 65.5] | 20.0 [4.3 to 92.0] | 24.6 [11.3 to 53.6] | 23.0 [11.1 to 47.8]
  B/Brisbane/60/2008 - Day 7 | 31.7 [15.0 to 67.3] | 56.6 [23.2 to 137.9] | 74.6 [32.7 to 170.3] | 80.0 [32.4 to 197.8]
  B/Brisbane/60/2008 - Day 21 | 40.0 [14.3 to 111.9] | 56.6 [20.8 to 154.2] | 121.3 [50.3 to 292.6] | 130.0 [57.7 to 292.5]
  B/Brisbane/60/2008 - Day 180 | 28.3 [9.4 to 85.2] | 35.6 [12.2 to 104.0] | 56.6 [24.2 to 132.5] | 56.6 [26.8 to 119.6]
  A/Perth/16/2009 (A/H3N2) - Day 0 | 56.6 [11.7 to 273.8] | 22.4 [6.4 to 78.6] | 37.3 [11.7 to 118.6] | 41.4 [12.4 to 138.3]
  A/Perth/16/2009 (A/H3N2) - Day 7 | 89.8 [23.6 to 341.1] | 89.8 [38.4 to 210.2] | 197.0 [75.0 to 517.1] | 139.3 [56.7 to 342.3]
  A/Perth/16/2009 (A/H3N2) - Day 21 | 89.8 [23.6 to 341.1] | 71.3 [24.4 to 207.9] | 211.1 [93.3 to 477.6] | 171.5 [83.6 to 351.8]
  A/Perth/16/2009 (A/H3N2) - Day 180 | 71.3 [15.1 to 337.3] | 35.6 [15.2 to 83.4] | 65.0 [24.8 to 170.6] | 74.6 [28.9 to 192.6]
  A/California/7/2009 (A/H1N1) - Day 0 | 10.0 [3.2 to 30.9] | 20.0 [2.8 to 140.8] | 32.5 [13.5 to 78.0] | 42.1 [17.6 to 101.0]
  A/California/7/2009 (A/H1N1) - Day 7 | 44.9 [14.0 to 144.0] | 142.5 [37.5 to 541.5] | 160.0 [68.9 to 371.7] | 242.5 [94.7 to 621.3]
  A/California/7/2009 (A/H1N1) - Day 21 | 50.4 [23.8 to 106.8] | 285.1 [41.8 to 1944.5] | 288.4 [88.6 to 939.2] | 242.5 [129.5 to 454.1]
  A/California/7/2009 (A/H1N1) - Day 180 | 15.9 [5.3 to 47.5] | 142.5 [32.3 to 629.2] | 91.9 [30.9 to 273.7] | 85.7 [45.3 to 162.3]

4. Secondary Outcome: Geometric Mean Titers (GMT) for Each of the Specific Influenza Strains Included in Vaccine Received by Participants in the 2012-2013 Season
Description: Blood was collected for HAI assay at Day 0 prior to vaccination and again at 7, 21 and 180 days following vaccination. The HAI assay was conducted with the three antigens in the 2012-2013 seasonal inactivated TIV. Within each 2012-2013 study arm, geometric mean titers and 95% confidence intervals were calculated for each antigen separately.
Time Frame: Days 0, 7, 21 and 180
Population: The analysis population includes all participants enrolled and vaccinated with the 2012-2013 vaccines who had blood collected at the visit. One RA Participant, Standard Dose and one Healthy Control, High Dose recipient are not included at Day 180 because the participant was out of window and lost to follow-up, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | RA Participants, 2012-2013 Fluzone Standard Dose | Healthy Controls, 2012-2013 Fluzone Standard Dose | RA Participants, 2012-2013 Fluzone High Dose | Healthy Controls, 2012-2013 Fluzone High Dose
Number analyzed (Participants) | 19 | 19 | 16 | 16
titers
  B/Wisconsin/1/2010 - Day 0 | 10.0 [6.3 to 15.8] | 9.6 [6.4 to 14.5] | 9.8 [6.7 to 14.4] | 7.1 [5.3 to 9.5]
  B/Wisconsin/1/2010 - Day 7 | 21.9 [12.4 to 38.7] | 11.8 [7.9 to 17.6] | 35.1 [21.1 to 58.4] | 19.6 [12.3 to 31.1]
  B/Wisconsin/1/2010 - Day 21 | 26.8 [16.1 to 44.6] | 14.4 [9.6 to 21.6] | 51.9 [32.3 to 83.4] | 20.0 [13.7 to 29.1]
  B/Wisconsin/1/2010 - Day 180 | 15.3 [8.6 to 27.1] | 10.8 [7.4 to 15.7] | 16.1 [10.1 to 25.7] | 9.1 [6.2 to 13.3]
  A/Victoria/361/2011 (A/H3N2) - Day 0 | 38.6 [19.7 to 75.4] | 38.6 [21.7 to 68.6] | 39.1 [16.6 to 92.5] | 45.6 [21.2 to 97.9]
  A/Victoria/361/2011 (A/H3N2) - Day 7 | 109.1 [62.7 to 189.8] | 97.8 [52.7 to 181.5] | 167.1 [75.7 to 368.8] | 226.3 [125.7 to 407.3]
  A/Victoria/361/2011 (A/H3N2) - Day 21 | 143.4 [81.0 to 253.8] | 113.1 [60.9 to 210.3] | 257.7 [136.9 to 484.9] | 252.2 [135.6 to 469.1]
  A/Victoria/361/2011 (A/H3N2) - Day 180 | 78.5 [39.7 to 155.0] | 59.8 [33.2 to 107.5] | 115.6 [58.8 to 227.3] | 100.8 [56.5 to 179.8]
  A/California/7/2009 (A/H1N1) - Day 0 | 31.8 [19.1 to 53.1] | 92.6 [50.6 to 169.2] | 35.1 [19.4 to 63.4] | 49.7 [20.6 to 119.9]
  A/California/7/2009 (A/H1N1) - Day 7 | 90.9 [52.2 to 158.3] | 148.7 [87.3 to 253.4] | 207.5 [81.6 to 527.6] | 203.0 [93.9 to 439.0]
  A/California/7/2009 (A/H1N1) - Day 21 | 120.6 [75.7 to 192.0] | 160.0 [88.8 to 288.4] | 442.9 [232.4 to 844.0] | 226.3 [109.8 to 466.3]
  A/California/7/2009 (A/H1N1) - Day 180 | 49.4 [28.3 to 86.4] | 117.3 [61.2 to 225.1] | 123.4 [55.8 to 272.8] | 96.2 [37.3 to 248.4]

5. Secondary Outcome: Number of Participants Reporting Solicited Systemic Symptoms Based on a Functional Grading Scale
Description: Participants maintained a memory aid to record daily the occurrence of systemic symptoms of feverishness, malaise, myalgia, headache, nausea, chills, arthralgia, shivering, and asthenia for 8 days after vaccination (Day 0-7) based on their interference with daily activities, with a severity grade of mild meaning no interference, moderate as some interference and severe as significant interference/prevented daily activity. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days.
Time Frame: Day 0 to Day 7
Population: The analysis population includes all participants enrolled and vaccinated in the study.
Measure: Number; unit: participants
Arm/Group | RA Participants, 2011-2012 Fluzone Standard Dose | Healthy Controls, 2011-2012 Fluzone Standard Dose | RA Participants, 2011-2012 Fluzone High Dose | Healthy Controls, 2011-2012 Fluzone High Dose | RA Participants, 2012-2013 Fluzone Standard Dose | Healthy Controls, 2012-2013 Fluzone Standard Dose | RA Participants, 2012-2013 Fluzone High Dose | Healthy Controls, 2012-2013 Fluzone High Dose
Number analyzed (Participants) | 6 | 6 | 10 | 10 | 19 | 19 | 16 | 16
participants
  Feverishness | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0
  Malaise | 1 | 0 | 5 | 1 | 13 | 3 | 13 | 1
  Myalgia | 2 | 0 | 4 | 1 | 14 | 2 | 13 | 2
  Headache | 4 | 1 | 3 | 5 | 8 | 5 | 8 | 2
  Nausea | 1 | 0 | 3 | 0 | 6 | 1 | 5 | 0
  Chills | 1 | 0 | 2 | 0 | 4 | 0 | 0 | 0
  Arthralgia | 6 | 0 | 7 | 0 | 18 | 1 | 14 | 2
  Shivering | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  Asthenia | 1 | 0 | 2 | 1 | 12 | 0 | 9 | 0

6. Secondary Outcome: Number of Participants Reporting Fever
Description: Participants were provided with a thermometer and a memory aid on which to record daily oral temperatures for 8 days after vaccination (Day 0-7). The protocol defined fever as oral temperature of 38.0 degrees Celsius or higher. Participants are counted as experiencing fever if they reported oral temperatures of 38.0 degrees Celsius or higher on any of the 8 days.
Time Frame: Day 0 to Day 7
Population: The analysis population includes all participants enrolled and vaccinated in the study.
Measure: Number; unit: participants
Arm/Group | RA Participants, 2011-2012 Fluzone Standard Dose | Healthy Controls, 2011-2012 Fluzone Standard Dose | RA Participants, 2011-2012 Fluzone High Dose | Healthy Controls, 2011-2012 Fluzone High Dose | RA Participants, 2012-2013 Fluzone Standard Dose | Healthy Controls, 2012-2013 Fluzone Standard Dose | RA Participants, 2012-2013 Fluzone High Dose | Healthy Controls, 2012-2013 Fluzone High Dose
Number analyzed (Participants) | 6 | 6 | 10 | 10 | 19 | 19 | 16 | 16
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Reporting Solicited Local Injection Site Reactions Based on a Functional Grading Scale
Description: Participants maintained a memory aid to record daily the occurrence of local injection site reactions of pain, tenderness, redness, and swelling for 8 days after vaccination (Day 0-7) based on their interference with daily activities, with a severity grade of mild meaning no interference, moderate as some interference and severe as significant interference/prevented daily activity. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days.
Time Frame: Day 0 to Day 7
Population: The analysis population includes all participants enrolled and vaccinated in the study.
Measure: Number; unit: participants
Arm/Group | RA Participants, 2011-2012 Fluzone Standard Dose | Healthy Controls, 2011-2012 Fluzone Standard Dose | RA Participants, 2011-2012 Fluzone High Dose | Healthy Controls, 2011-2012 Fluzone High Dose | RA Participants, 2012-2013 Fluzone Standard Dose | Healthy Controls, 2012-2013 Fluzone Standard Dose | RA Participants, 2012-2013 Fluzone High Dose | Healthy Controls, 2012-2013 Fluzone High Dose
Number analyzed (Participants) | 6 | 6 | 10 | 10 | 19 | 19 | 16 | 16
participants
  Pain | 0 | 3 | 1 | 4 | 4 | 6 | 8 | 5
  Tenderness | 5 | 5 | 6 | 9 | 6 | 12 | 12 | 10
  Redness | 0 | 0 | 0 | 1 | 1 | 3 | 5 | 2
  Swelling | 1 | 0 | 1 | 0 | 3 | 6 | 5 | 6

8. Secondary Outcome: Number of Participants Reporting Solicited Quantitative Local Injection Site Reactions
Description: Participants maintained a memory aid to record daily the occurrence of local reactions of redness and swelling for 8 days after vaccination (Day 0-7). If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they reported experiencing the reaction with any measurement greater than 0 mm on any of the 8 days.
Time Frame: Day 0 to Day 7
Population: The analysis population includes all participants enrolled and vaccinated in the study.
Measure: Number; unit: participants
Arm/Group | RA Participants, 2011-2012 Fluzone Standard Dose | Healthy Controls, 2011-2012 Fluzone Standard Dose | RA Participants, 2011-2012 Fluzone High Dose | Healthy Controls, 2011-2012 Fluzone High Dose | RA Participants, 2012-2013 Fluzone Standard Dose | Healthy Controls, 2012-2013 Fluzone Standard Dose | RA Participants, 2012-2013 Fluzone High Dose | Healthy Controls, 2012-2013 Fluzone High Dose
Number analyzed (Participants) | 6 | 6 | 10 | 10 | 19 | 19 | 16 | 16
participants
  Redness | 0 | 0 | 0 | 1 | 1 | 3 | 5 | 2
  Swelling | 1 | 0 | 1 | 0 | 3 | 6 | 5 | 6

9. Primary Outcome: Number of RA Participants in the 2012-2013 Season Who Achieved Seroconversion at Day 21 Against Each of the 3 Specific Influenza Strains in Vaccine the Participant Received
Description: Blood was collected from RA participants prior to vaccination and at the 21 day follow up visit for testing in the HAI assay with 2012-2013 seasonal influenza vaccine strains virus as the assay antigens. A participant met the threshold of seroconversion if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to and Day 21 following immunization
Population: The analysis population includes all RA participants enrolled and vaccinated with the 2012-2013 vaccines.
Measure: Number; unit: participants
Arm/Group | RA Participants, 2012-2013 Fluzone Standard Dose | RA Participants, 2012-2013 Fluzone High Dose
Number analyzed (Participants) | 19 | 16
participants
  B/Wisconsin/1/2010 | 6 | 9
  A/Victoria/361/2011 (A/H3N2) | 9 | 10
  A/California/7/2009 (A/H1N1) | 8 | 12
Statistical Analysis 1: Comparison: RA Participants, 2012-2013 Fluzone Standard Dose vs RA Participants, 2012-2013 Fluzone High Dose; This is the comparison for the B/Wisconsin/1/2010 strain; Test type: Superiority or Other; p = 0.182, Fisher Exact
Statistical Analysis 2: Comparison: RA Participants, 2012-2013 Fluzone Standard Dose vs RA Participants, 2012-2013 Fluzone High Dose; This is the comparison for the A/Victoria/361/2011 (A/H3N2) strain; Test type: Superiority or Other; p = 0.500, Fisher Exact
Statistical Analysis 3: Comparison: RA Participants, 2012-2013 Fluzone Standard Dose vs RA Participants, 2012-2013 Fluzone High Dose; This is the comparison for the A/California/7/2009 (A/H1N1) strain; Test type: Superiority or Other; p = 0.087, Fisher Exact

10. Secondary Outcome: Number of RA Participants in the 2011-2012 Season Who Achieved Seroconversion at Days 7 and 180 Against Each of the 3 Specific Influenza Strains in Vaccine the Participant Received
Description: Blood was collected from RA participants prior to vaccination and at the Days 7 and 180 follow up visits for testing in the HAI assay with 2011-2012 seasonal influenza vaccine strains virus as the assay antigens. A participant met the threshold of seroconversion if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to and Days 7 and 180 following immunization
Population: The analysis population includes all RA subjects enrolled and vaccinated with the 2011-2012 vaccines.
Measure: Number; unit: participants
Arm/Group | RA Participants, 2011-2012 Fluzone Standard Dose | RA Participants, 2011-2012 Fluzone High Dose
Number analyzed (Participants) | 6 | 10
participants
  B/Brisbane/60/2008 - Day 7 | 0 | 4
  B/Brisbane/60/2008 - Day 180 | 0 | 3
  A/Perth/16/2009 (A/H3N2) - Day 7 | 1 | 6
  A/Perth/16/2009 (A/H3N2) - Day 180 | 0 | 2
  A/California/7/2009 (A/H1N1) - Day 7 | 3 | 6
  A/California/7/2009 (A/H1N1) - Day 180 | 0 | 2
Statistical Analysis 1: Comparison: RA Participants, 2011-2012 Fluzone Standard Dose vs RA Participants, 2011-2012 Fluzone High Dose; This is the comparison for the B/Brisbane/60/2008 strain at Day 7; Test type: Superiority or Other; p = 0.234, Fisher Exact
Statistical Analysis 2: Comparison: RA Participants, 2011-2012 Fluzone Standard Dose vs RA Participants, 2011-2012 Fluzone High Dose; This is the comparison for the B/Brisbane/60/2008 strain at Day 180; Test type: Superiority or Other; p = 0.250, Fisher Exact
Statistical Analysis 3: Comparison: RA Participants, 2011-2012 Fluzone Standard Dose vs RA Participants, 2011-2012 Fluzone High Dose; This is the comparison for the A/Perth/16/2009 (A/H3N2) strain at Day 7; Test type: Superiority or Other; p = 0.145, Fisher Exact
Statistical Analysis 4: Comparison: RA Participants, 2011-2012 Fluzone Standard Dose vs RA Participants, 2011-2012 Fluzone High Dose; This is the comparison for the A/Perth/16/2009 (A/H3N2) strain at Day 180; Test type: Superiority or Other; p = 0.500, Fisher Exact
Statistical Analysis 5: Comparison: RA Participants, 2011-2012 Fluzone Standard Dose vs RA Participants, 2011-2012 Fluzone High Dose; This is the comparison for the A/California/7/2009 (A/H1N1) strain at Day 7; Test type: Superiority or Other; p = 0.999, Fisher Exact
Statistical Analysis 6: Comparison: RA Participants, 2011-2012 Fluzone Standard Dose vs RA Participants, 2011-2012 Fluzone High Dose; This is the comparison for the A/California/7/2009 (A/H1N1) strain at Day 180; Test type: Superiority or Other; p = 0.500, Fisher Exact

11. Secondary Outcome: Number of RA Participants in the 2012-2013 Season Who Achieved Seroconversion at Days 7 and 180 Against Each of the 3 Specific Influenza Strains in Vaccine the Participant Received
Description: Blood was collected from RA participants prior to vaccination and at the Days 7 and 180 follow up visits for testing in the HAI assay with 2012-2013 seasonal influenza vaccine strains virus as the assay antigens. A participant met the threshold of seroconversion if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to and Days 7 and 180 following immunization
Population: The analysis population includes RA participants enrolled and vaccinated with the 2012-2013 vaccines who had blood collected at the visit. One RA Participant, Standard Dose recipient is not included at Day 180 because the participant was out of window.
Measure: Number; unit: participants
Arm/Group | RA Participants, 2012-2013 Fluzone Standard Dose | RA Participants, 2012-2013 Fluzone High Dose
Number analyzed (Participants) | 19 | 16
participants
  B/Wisconsin/1/2010 - Day 7 | 5 | 6
  B/Wisconsin/1/2010 - Day 180 | 2 | 2
  A/Victoria/361/2011 (A/H3N2) - Day 7 | 6 | 7
  A/Victoria/361/2011 (A/H3N2) - Day 180 | 5 | 7
  A/California/7/2009 (A/H1N1) - Day 7 | 6 | 9
  A/California/7/2009 (A/H1N1) - Day 180 | 1 | 7
Statistical Analysis 1: Comparison: RA Participants, 2012-2013 Fluzone Standard Dose vs RA Participants, 2012-2013 Fluzone High Dose; This is the comparison for the B/Wisconsin/1/2010 strain at Day 7; Test type: Superiority or Other; p = 0.716, Fisher Exact
Statistical Analysis 2: Comparison: RA Participants, 2012-2013 Fluzone Standard Dose vs RA Participants, 2012-2013 Fluzone High Dose; This is the comparison for the B/Wisconsin/1/2010 strain at Day 180; Test type: Superiority or Other; p = 0.999, Fisher Exact
Statistical Analysis 3: Comparison: RA Participants, 2012-2013 Fluzone Standard Dose vs RA Participants, 2012-2013 Fluzone High Dose; This is the comparison for the A/Victoria/361/2011 (A/H3N2) strain at Day 7; Test type: Superiority or Other; p = 0.503, Fisher Exact
Statistical Analysis 4: Comparison: RA Participants, 2012-2013 Fluzone Standard Dose vs RA Participants, 2012-2013 Fluzone High Dose; This is the comparison for the A/Victoria/361/2011 (A/H3N2) strain at Day 180; Test type: Superiority or Other; p = 0.475, Fisher Exact
Statistical Analysis 5: Comparison: RA Participants, 2012-2013 Fluzone Standard Dose vs RA Participants, 2012-2013 Fluzone High Dose; This is the comparison for the A/California/7/2009 (A/H1N1) strain at Day 7; Test type: Superiority or Other; p = 0.182, Fisher Exact
Statistical Analysis 6: Comparison: RA Participants, 2012-2013 Fluzone Standard Dose vs RA Participants, 2012-2013 Fluzone High Dose; This is the comparison for the A/California/7/2009 (A/H1N1) strain at Day 180; Test type: Superiority or Other; p = 0.014, Fisher Exact

12. Secondary Outcome: Number of RA Participants With a Worsening Rheumatoid Arthritis Status During the Course of the Study, Based on the RAPID3 Score From the NP2 Questionnaire
Description: The RAPID 3 score is an index of the three patient-reported measures from the Multi-Dimensional Health Assessment Questionnaire (MDHAQ) R808 and serves as an assessment of patient status for those with rheumatoid arthritis. The score consists of the cumulative total of the Function (FN), Pain (PN), and Patient Global (PTGL) values. The severity of the RAPID 3 score is categorized as: >12=High Severity; 6.1-12=Moderate Severity; 3.1-6=Low Severity; and ≤3=Remission. The NP2 questionnaire was completed by RA participants at all clinic visits. Scores at Days 7, 21 and 180 were compared to Day 0 to determine worsening, defined as moving from the baseline category to a more severe category.
Time Frame: Day 0 to Days 7, 21 and 180
Population: All RA participants are included in the analysis population for this outcome measure.
Measure: Number; unit: participants
Arm/Group | RA Participants, 2011-2012 Fluzone Standard Dose | RA Participants, 2011-2012 Fluzone High Dose | RA Participants, 2012-2013 Fluzone Standard Dose | RA Participants, 2012-2013 Fluzone High Dose
Number analyzed (Participants) | 6 | 10 | 19 | 16
participants
  Day 7 | 0 | 0 | 2 | 2
  Day 21 | 1 | 2 | 2 | 2
  Day 180 | 0 | 3 | 3 | 3

13. Secondary Outcome: Number of Participants in the 2011-2012 Season Who Achieved Seroconversion at Days 7, 21 and 180 Against Each of the 3 Specific Influenza Strains in Vaccine the Participant Received
Description: Blood was collected from all participants prior to vaccination and at the Days 7, 21 and 180 follow up visits for testing in the HAI assay with 2011-2012 seasonal influenza vaccine strains virus as the assay antigens. A participant met the threshold of seroconversion if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to and Days 7, 21 and 180 following immunization
Population: The analysis population includes all subjects enrolled and vaccinated with the 2011-2012 vaccines.
Measure: Number; unit: participants
Arm/Group | RA Participants, 2011-2012 Fluzone Standard Dose | Healthy Controls, 2011-2012 Fluzone Standard Dose | RA Participants, 2011-2012 Fluzone High Dose | Healthy Controls, 2011-2012 Fluzone High Dose
Number analyzed (Participants) | 6 | 6 | 10 | 10
participants
  B/Brisbane/60/2008 - Day 7 | 0 | 2 | 4 | 4
  B/Brisbane/60/2008 - Day 21 | 1 | 3 | 6 | 5
  B/Brisbane/60/2008 - Day 180 | 0 | 1 | 3 | 3
  A/Perth/16/2009 (A/H3N2) - Day 7 | 1 | 2 | 6 | 5
  A/Perth/16/2009 (A/H3N2) - Day 21 | 1 | 2 | 6 | 6
  A/Perth/16/2009 (A/H3N2) - Day 180 | 0 | 1 | 2 | 2
  A/California/7/2009 (A/H1N1) - Day 7 | 3 | 4 | 6 | 5
  A/California/7/2009 (A/H1N1) - Day 21 | 4 | 4 | 7 | 6
  A/California/7/2009 (A/H1N1) - Day 180 | 0 | 3 | 2 | 2
Statistical Analysis 1: Comparison: RA Participants, 2011-2012 Fluzone Standard Dose vs Healthy Controls, 2011-2012 Fluzone Standard Dose; This is the comparison for the B/Brisbane/60/2008 strain at Day 21; Test type: Superiority or Other; p = 0.317, McNemar
Statistical Analysis 2: Comparison: RA Participants, 2011-2012 Fluzone Standard Dose vs Healthy Controls, 2011-2012 Fluzone Standard Dose; This is the comparison for the A/Perth/16/2009 (A/H3N2) strain at Day 21; Test type: Superiority or Other; p = 0.564, McNemar
Statistical Analysis 3: Comparison: RA Participants, 2011-2012 Fluzone Standard Dose vs Healthy Controls, 2011-2012 Fluzone Standard Dose; This is the comparison for the A/California/7/2009 (A/H1N1) strain at Day 21; Test type: Superiority or Other; p = 0.999, McNemar
Statistical Analysis 4: Comparison: RA Participants, 2011-2012 Fluzone High Dose vs Healthy Controls, 2011-2012 Fluzone High Dose; This is the comparison for the B/Brisbane/60/2008 strain at Day 21; Test type: Superiority or Other; p = 0.564, McNemar
Statistical Analysis 5: Comparison: RA Participants, 2011-2012 Fluzone High Dose vs Healthy Controls, 2011-2012 Fluzone High Dose; This is the comparison for the A/Perth/16/2009 (A/H3N2) strain at Day 21; Test type: Superiority or Other; p = 0.999, McNemar
Statistical Analysis 6: Comparison: RA Participants, 2011-2012 Fluzone High Dose vs Healthy Controls, 2011-2012 Fluzone High Dose; This is the comparison for the A/California/7/2009 (A/H1N1) strain at Day 21; Test type: Superiority or Other; p = 0.655, McNemar

14. Secondary Outcome: Number of Participants in the 2012-2013 Season Who Achieved Seroconversion at Days 7, 21 and 180 Against Each of the 3 Specific Influenza Strains in Vaccine the Participant Received
Description: Blood was collected from all participants prior to vaccination and at the Days 7, 21 and 180 follow up visits for testing in the HAI assay with 2012-2013 seasonal influenza vaccine strains virus as the assay antigens. A participant met the threshold of seroconversion if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to and Days 7, 21 and 180 following immunization
Population: The analysis population includes all subjects enrolled and vaccinated with the 2012-2013 vaccines who had blood collected at the visit. One RA Participant, Standard Dose and one Healthy Control, High Dose recipient are not included at Day 180 because the participant was out of window and lost to follow-up, respectively.
Measure: Number; unit: participants
Arm/Group | RA Participants, 2012-2013 Fluzone Standard Dose | Healthy Controls, 2012-2013 Fluzone Standard Dose | RA Participants, 2012-2013 Fluzone High Dose | Healthy Controls, 2012-2013 Fluzone High Dose
Number analyzed (Participants) | 19 | 19 | 16 | 16
participants
  B/Wisconsin/1/2010 - Day 7 | 5 | 0 | 6 | 5
  B/Wisconsin/1/2010 - Day 21 | 6 | 3 | 9 | 5
  B/Wisconsin/1/2010 - Day 180 | 2 | 1 | 2 | 0
  A/Victoria/361/2011 (A/H3N2) - Day 7 | 6 | 6 | 7 | 9
  A/Victoria/361/2011 (A/H3N2) - Day 21 | 9 | 8 | 10 | 11
  A/Victoria/361/2011 (A/H3N2) - Day 180 | 5 | 2 | 7 | 4
  A/California/7/2009 (A/H1N1) - Day 7 | 6 | 1 | 9 | 7
  A/California/7/2009 (A/H1N1) - Day 21 | 8 | 3 | 12 | 7
  A/California/7/2009 (A/H1N1) - Day 180 | 1 | 2 | 7 | 1
Statistical Analysis 1: Comparison: RA Participants, 2012-2013 Fluzone Standard Dose vs Healthy Controls, 2012-2013 Fluzone Standard Dose; This is the comparison for the B/Wisconsin/1/2010 strain at Day 21; Test type: Superiority or Other; p = 0.180, McNemar
Statistical Analysis 2: Comparison: RA Participants, 2012-2013 Fluzone Standard Dose vs Healthy Controls, 2012-2013 Fluzone Standard Dose; This is the comparison for the A/Victoria/361/2011 (A/H3N2) strain at Day 21; Test type: Superiority or Other; p = 0.763, McNemar
Statistical Analysis 3: Comparison: RA Participants, 2012-2013 Fluzone Standard Dose vs Healthy Controls, 2012-2013 Fluzone Standard Dose; This is the comparison for the A/California/7/2009 (A/H1N1) strain at Day 21; Test type: Superiority or Other; p = 0.096, McNemar
Statistical Analysis 4: Comparison: RA Participants, 2012-2013 Fluzone High Dose vs Healthy Controls, 2012-2013 Fluzone High Dose; This is the comparison for the B/Wisconsin/1/2010 strain at Day 21; Test type: Superiority or Other; p = 0.157, McNemar
Statistical Analysis 5: Comparison: RA Participants, 2012-2013 Fluzone High Dose vs Healthy Controls, 2012-2013 Fluzone High Dose; This is the comparison for the A/Victoria/361/2011 (A/H3N2) strain at Day 21; Test type: Superiority or Other; p = 0.705, McNemar
Statistical Analysis 6: Comparison: RA Participants, 2012-2013 Fluzone High Dose vs Healthy Controls, 2012-2013 Fluzone High Dose; This is the comparison for the A/California/7/2009 (A/H1N1) strain at Day 21; Test type: Superiority or Other; p = 0.132, McNemar

ADVERSE EVENTS:
Time Frame: Solicited events were collected for 8 days after vaccination, unsolicited non-serious adverse events through 21 days after vaccination, and serious adverse events and new onset chronic medical conditions through 180 days after vaccination.
Description: For events solicited on a Memory Aid in the 8 days after vaccination, a participant was considered to have one event if it was reported as experienced at any time in the 8 day period.
Arm/Group | RA Participants, 2011-2012 Fluzone Standard Dose | Healthy Controls, 2011-2012 Fluzone Standard Dose | RA Participants, 2011-2012 Fluzone High Dose | Healthy Controls, 2011-2012 Fluzone High Dose | RA Participants, 2012-2013 Fluzone Standard Dose | Healthy Controls, 2012-2013 Fluzone Standard Dose | RA Participants, 2012-2013 Fluzone High Dose | Healthy Controls, 2012-2013 Fluzone High Dose
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/10 | 0/10 | 1/19 | 0/19 | 0/16 | 1/16
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 10/10 | 9/10 | 18/19 | 14/19 | 16/16 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RA Participants, 2011-2012 Fluzone Standard Dose (N=6) | Healthy Controls, 2011-2012 Fluzone Standard Dose (N=6) | RA Participants, 2011-2012 Fluzone High Dose (N=10) | Healthy Controls, 2011-2012 Fluzone High Dose (N=10) | RA Participants, 2012-2013 Fluzone Standard Dose (N=19) | Healthy Controls, 2012-2013 Fluzone Standard Dose (N=19) | RA Participants, 2012-2013 Fluzone High Dose (N=16) | Healthy Controls, 2012-2013 Fluzone High Dose (N=16)
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RA Participants, 2011-2012 Fluzone Standard Dose (N=6) | Healthy Controls, 2011-2012 Fluzone Standard Dose (N=6) | RA Participants, 2011-2012 Fluzone High Dose (N=10) | Healthy Controls, 2011-2012 Fluzone High Dose (N=10) | RA Participants, 2012-2013 Fluzone Standard Dose (N=19) | Healthy Controls, 2012-2013 Fluzone Standard Dose (N=19) | RA Participants, 2012-2013 Fluzone High Dose (N=16) | Healthy Controls, 2012-2013 Fluzone High Dose (N=16)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Solicited as "feverishness" on the memory aid
Malaise (General disorders) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 13 (13) | 3 (3) | 13 (13) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 14 (14) | 2 (2) | 13 (13) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 1 (1) | 3 (3) | 5 (5) | 8 (8) | 5 (5) | 8 (8) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 6 (6) | 1 (1) | 5 (5) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) — Solicited as "chills" on the memory aid
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) — Solicited as "shivering" on the memory aid
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 7 (7) | 0 (0) | 18 (18) | 1 (1) | 14 (14) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 12 (12) | 0 (0) | 9 (9) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 4 (4) | 6 (6) | 8 (8) | 5 (5)
Tenderness (General disorders) | 5 (5) | 5 (5) | 6 (6) | 9 (9) | 6 (6) | 12 (12) | 12 (12) | 10 (10)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 5 (5) | 2 (2)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 6 (6) | 5 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less